CLINICAL TRIAL: NCT00254410
Title: Phase 2 Study of the Activity and Safety of Fludarabine, Cyclophosphamide, and Mitoxantrone Plus Rituximab (FCM-R) With Pegfilgrastim (Neulasta) as Frontline Therapy for Patients < 70 Years With Chronic Lymphocytic Leukemia
Brief Title: FCM-R (Fludarabine, Cyclophosphamide, Mitoxantrone, Rituximab) in Previously Untreated Patients With Chronic Lymphocytic Leukemia (CLL) < 70 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0106; NCI-2010-00437 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Untreated; Fludarabine; Fludara; Cyclophosphamide; Cytoxan; Mitoxantrone; Novantrone; Rituximab; Rituxan; Pegylated Filgrastim; Neupogen
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mitoxantrone; Rituximab; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FCM-R + Pegylated Filgrastim (Experimental): Fludarabine 25 mg/m2 on Days 2,3,4 i.v. 5-30 mins for course 1, and on Days 1 - 3 for courses 2 - 6. Cyclophosphamide 250 mg/m2 on Day 2,3,4 i.v. 5-30 mins for course 1, and on Days1 - 3 for courses 2 - 6. Mitoxantrone 6 mg/m2 on Day 2 i.v. 30-60 mins for course 1, and on Day 1 for courses 2 - 6. Rituximab 375 mg/m2 on Day 1 i.v. 2-6 hours for course 1 and 500 mg/m2 on Day 1 for courses 2 - 6. Pegylated Filgrastim - 6 mg on Day 4,s.c. for course 1 and on Day 3 for courses 2 - 6.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mitoxantrone; Drug: Rituximab; Drug: Filgrastim

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25 mg/m2 on Days 2,3,4 i.v. 5-30 mins for course 1, and on Days 1 - 3 for courses 2 - 6
  Other Names: Fludara®
Drug: Cyclophosphamide — Cyclophosphamide 250 mg/m2 on Day 2,3,4 i.v. 5-30 mins for course 1, and on Days1 - 3 for courses 2 - 6.
  Other Names: Cytoxan®
Drug: Mitoxantrone — Mitoxantrone 6 mg/m2 on Day 2 i.v. 30-60 mins for course 1, and on Day 1 for courses 2 - 6.
  Other Names: Novantrone®
Drug: Rituximab — Rituximab 375 mg/m2 on Day 1 i.v. 2-6 hours for course 1 and 500 mg/m2 on Day 1 for courses 2 - 6.
  Other Names: Rituxan®
Drug: Filgrastim — Pegylated Filgrastim - 6 mg on Day 4,s.c. for course 1 and on Day 3 for courses 2 - 6.
  Other Names: Neupogen®

SUMMARY:
The goal of this clinical research study is to learn if using a combination of fludarabine, cyclophosphamide, and mitoxantrone plus rituximab, with the growth factor pegylated filgrastim, will improve the response to treatment, and increase the time this response lasts, for patients with previously untreated CLL. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Fludarabine, cyclophosphamide, and mitoxantrone are chemotherapy drugs that are used in the treatment of CLL. Rituximab is a monoclonal antibody that binds to CLL cells and causes cell death. Pegfilgrastim (Neulasta) is a growth factor that helps the bone marrow to produce white cells (neutrophils) and is an approved drug to treat the suppression of marrow function caused by chemotherapy.

If you are eligible to take part in the study, you will begin treatment. Rituximab will be given through a needle in your vein (IV) on Day 1 of Courses 1-6. The first infusion may take up to 8 hours. For every dose of rituximab after that, the infusion may take 2-4 hours. The length of the infusion time depends on whether you have any reactions to the infusion. The dose level of rituximab may be increased for Cycles 2-6 as well. The drugs acetaminophen (Tylenol) and diphenhydramine hydrochloride (Benadryl) will be given before each dose of rituximab. This will be done to decrease the risk of side effects. If side effects do occur during rituximab treatment, the drug may have to be stopped until the side effects go away and then restarted, so your time in the outpatient area may be longer if that occurs.

One day after the first dose of rituximab (Day 2), fludarabine and cyclophosphamide will be given by IV every day for 3 days (Days 2, 3, and 4), and mitoxantrone will be given by IV on Day 2. Fludarabine and cyclophosphamide will be given as 30-minute infusions, while the infusion of mitoxantrone will take 30-60 minutes. After the first treatment cycle, all the drugs will be given on Days 1, 2, and 3 for every cycle after that. Pegfilgrastim will be given as a subcutaneous injection (an injection under the skin) once per treatment cycle, right after you receive the last chemotherapy drug (in other words, on Day 4 during the first cycle, and on Day 3 for every cycle after that). Other IV fluids, such as saline, will be given on all of the treatment days to keep you hydrated, which means that each clinic visit will take about 6 hours. The combination will be repeated once every 4 to 6 weeks for a total of 6 courses.

The first treatment will be given at the University of Texas MD Anderson Cancer Center (UTMDACC) outpatient clinic. The other 5 courses can be performed either at UTMDACC or at home with your regular physician.

During each treatment cycle, you will have blood samples (about 1 teaspoon each) drawn once every 1-2 weeks. Bone marrow biopsies will be performed at the end of Cycles 3 and 6 of chemotherapy.

With the exception of rituximab, the same doses of all other drugs will be used throughout the study unless side effects become severe. In that case, the dose may be lowered or the treatment may be stopped. You will be taken off study if the disease gets worse.

After Course 6 of chemotherapy is finished, you will have blood tests (about 2 teaspoons each) performed every 6-12 months.

This is an investigational study. The FDA has approved all of the drugs used in this study, and they are commercially available. However, their use in this study and in this combination is considered investigational. Up to 30 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated CLL, CLL/ prolymphocytic leukemia (PLL), or small lymphocytic lymphoma (SLL) with indication for therapy (Indications for therapy include at least one of the following: i) one or more disease-related symptoms [fever, night sweats, weight loss, pronounced fatigue]; ii) advanced stage disease (Rai stage >/= 3 or Binet stage C); iii) autoimmune anemia and/or thrombocytopenia that is unresponsive to other therapies; iv) massive or progressive hepatomegaly and/or splenomegaly and/or lymphadenopathy; iv) recurrent infections; v) rapid lymphocyte doubling time of < 6 months).
2. Age < 70 years.
3. Adequate liver function (total bilirubin </= 2.5 mg/dL, serum glutamate pyruvate transaminase (SGPT) </=4 x ULN) and renal function (serum creatinine </= 2.0 mg/dL). Patients with renal or liver dysfunction due to suspected organ infiltration by lymphocytes may be eligible after discussion with the Principal Investigator, but upper limits for creatinine even under these circumstances must be creatinine < 3mg/dL and bilirubin < 6 mg/dL. Patients with Gilbert's syndrome may be entered on study with bilirubin levels </= 4 mg/dL.
4. Beta-2-microglobulin </= 4 mg/dL.
5. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
6. Signed informed consent in keeping with the policies of the hospital.
7. Male and female patients who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc) to avoid pregnancy. Female patients of childbearing potential (non-childbearing is defined as >/= 1 year postmenopausal or surgically sterilized) need a negative serum or urine pregnancy test within 14 days of study enrollment.

Exclusion Criteria:

1. Active hepatitis B (at least one of the following markers positive: HBsAg, HBeAg, Immunoglobulin M (IgM) hepatitis B core antibody (anti-HBc), Hepatitis B (HBV) DNA).
2. Concurrent chemotherapy or immunotherapy.
3. Pregnant patients.
4. History of HIV
5. Symptomatic central nervous system (CNS) disease
6. Symptomatic heart disease (NYHA class >/= 3) or left ventricle (LV) ejection fraction < 40% (by multiple gated acquisition scan (MUGA) or echocardiogram)

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03-14 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PHD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2005 to April 2006. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | FCM-R + Pegylated Filgrastim
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FCM-R + Pegylated Filgrastim
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate at 3 Months
Description: Clinical Response Rate (combined morphological [NCI Working Group (WG) criteria] + flow cytometry criteria) at 3 months following treatment. Courses will be repeated every 28 to 42 days (+/- 7 days) depending on recovery of peripheral blood counts and toxicities for a maximum of 6 courses. Patients will be evaluated for response after 3 and 6 courses. Bone marrow biopsies will be performed at the end of Cycles 3 and 6 of chemotherapy.
Time Frame: End of cycle 3
Measure: Count of Participants; unit: Participants
Arm/Group | FCM-R + Pegylated Filgrastim
Number analyzed (Participants) | 30
Participants | 29

2. Primary Outcome: Clinical Response Rate at 6 Months
Description: Clinical Response Rate (combined morphological [NCI WG criteria] + flow cytometry criteria) at 6 months following treatment. Courses will be repeated every 28 to 42 days (+/- 7 days) depending on recovery of peripheral blood counts and toxicities for a maximum of 6 courses. Patients will be evaluated for response after 3 and 6 courses. Bone marrow biopsies will be performed at the end of Cycles 3 and 6 of chemotherapy.
Time Frame: End of Cycle 6
Population: One participant showed progression while on therapy and was taken off study after 3 courses. Of the 30 participants who started therapy, one participant was not analyzed at the end of cycle 6.
Measure: Count of Participants; unit: Participants
Arm/Group | FCM-R + Pegylated Filgrastim
Number analyzed (Participants) | 29
Participants | 28

3. Secondary Outcome: Molecular Response Rate at 3 Months
Description: Molecular response rate (PCR for immunoglobulin heavy chain (IgH) rearrangements) at 3 months following treatment. Courses will be repeated every 28 to 42 days (+/- 7 days) depending on recovery of peripheral blood counts and toxicities for a maximum of 6 courses. Patients will be evaluated for response after 3 and 6 courses. Bone marrow biopsies will be performed at the end of Cycles 3 and 6 of chemotherapy.
Time Frame: End of cycle 3
Measure: Count of Participants; unit: Participants
Arm/Group | FCM-R + Pegylated Filgrastim
Number analyzed (Participants) | 30
Participants | 17

4. Secondary Outcome: Molecular Response Rate at 6 Months
Description: Molecular response rate (PCR for IgH rearrangements) at 6 months following treatment. Courses will be repeated every 28 to 42 days (+/- 7 days) depending on recovery of peripheral blood counts and toxicities for a maximum of 6 courses. Patients will be evaluated for response after 3 and 6 courses. Bone marrow biopsies will be performed at the end of Cycles 3 and 6 of chemotherapy.
Time Frame: End of 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | FCM-R + Pegylated Filgrastim
Number analyzed (Participants) | 29
Participants | 10

ADVERSE EVENTS:
Time Frame: Up to 10 months
Arm/Group | FCM-R + Pegylated Filgrastim
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCM-R + Pegylated Filgrastim (N=30)
Fever (General disorders) | 2 (2)
Neutropenic Fever (Infections and infestations) | 3 (3)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCM-R + Pegylated Filgrastim (N=30)
Neutropenia (Blood and lymphatic system disorders) | 26 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (24)
Anemia (Blood and lymphatic system disorders) | 23 (23)
Nausea (Gastrointestinal disorders) | 23 (23)
Fatigue (General disorders) | 18 (18)
Fever (General disorders) | 16 (16)
Neutropenic Fever (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Chills (General disorders) | 6 (6)
Sweats (General disorders) | 6 (6)
Upper Respiratory Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Indigestion (Gastrointestinal disorders) | 4 (4)
Joint/Bone Pain (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Body Aches (General disorders) | 3 (3)
Weakness (General disorders) | 2 (2)
Autoimmune hemolytic anemia (AIHA) (Immune system disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT00254410/Prot_SAP_000.pdf